CLINICAL TRIAL: NCT00122798
Title: Improved Stroke Outcome at 6 Months Attained by a Chain of Structured Acute Treatment With Integrated Rehabilitation and Supported Discharge
Brief Title: Improved Stroke Outcome at 6 Months
Status: Completed | Type: Observational
Sponsor: Kantonsspital Baden (Other)
Collaborators: RehaClinic Zurzach (Unknown)
Other Study IDs: EK 50
Record Dates: First submitted 2005-07-21; First posted 2005-07-22 (Estimated); Last update posted 2006-06-27 (Estimated); Status verified 2004-12

CONDITIONS: Stroke
Keywords: Stroke, stroke treatment, atrial fibrillation, medication, rehabilitation
MeSH Terms: conditions — Stroke; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Stroke treatment

SUMMARY:
The investigators implemented a structured chain of acute stroke care with early integrated rehabilitation. The mortality at 6 months was lower (12%) compared to 23% in the International Stroke Trial (IST) and 39% (67%) of the patients were dead or dependent, which is superior compared to international data.

DETAILED DESCRIPTION:
Background/Aim of the study: To further reduce the 6 months stroke morbidity and mortality in a high volume stroke hospital and to compare the results with national and international data.

Methods: 204 consecutive stroke patients are analyzed in a prospective study in a single center teaching institution. The intervention consists of a structured therapeutic chain of 290 collaborating GPs, a standardised acute hospital proceeding overlapping with an early integrated neurovascular rehabilitation within the same institution. Primary endpoints include death and dependence at 6 months, secondary endpoints are the length of hospital stay (LOS) and the quantitative analysis of physical and psychosocial impairments. The data are directly compared with the same endpoints of the Swiss subgroup of the international stroke trial (IST) and recent international data.

Results: At 6 months, mortality is significantly lower with 12 % (compared to 23 % in the IST trial) and only 39 % (67 %) of the patients are dead or dependent. Stroke severity is similar as in other study populations. Median LOS is 15 days in the acute clinic and 39 days in the rehabilitation institution. The psychosocial outcome compares favorably to a matched control group.

Conclusions: A structured chain of acute stroke treatment overlapping with an early integrated rehabilitation is superior compared to national and international ischemic stroke trial data.

ELIGIBILITY:
Inclusion Criteria:

* An acute cerebrovascular event (ischemic stroke or intra-cerebral bleeding (ICB)) with the signs and symptoms of an acute stroke according to the World Health Organisation definition of acute stroke within the last 12 hours without the need or possibility of a neurosurgical intervention;
* No thrombolytic therapy within the first 3 hours (in order to allow the correct comparison with the Swiss cohort of the IST trial)
* The informed consent of the patient or, if not possible, of the next of kindred
* Living at home before the event
* Lack of participation in another trial

Exclusion Criteria:

* Transient ischemic attack (TIA) resp. full recovery within 24 hours after the event

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2002-01; Study Completion 2005-01

CONTACTS AND LOCATIONS:
Overall Officials: Juerg H Beer, M.D, Principal Investigator — Dept of Medicine, Kantonsspital Baden, Switzerland
Locations (1):
- Kantonsspital Baden, Baden, Canton of Aargau, Switzerland

REFERENCES:
- See also: Related Info — http://www.ksb.ch